CLINICAL TRIAL: NCT03922230
Title: Digestive Tract Tumor Research Based on ctDNA Methylation Detection Technology and Early Non-invasive Screening: Exploration and Verification of DNA Methylolation in Early Screening of Esophageal Cancer
Brief Title: Exploration and Verification of DNA Methylolation in Early Screening of Esophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2019-015
Record Dates: First submitted 2019-03-15; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cancer; DNA methylolation; early screening
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early esophageal cancer group: Pathological examination diagnosed as Early esophageal cancer.The ratio of male to female is 3:1, and the age is between 50 and 70 years old.
- Middle and advanced ES group: Pathological examination diagnosed as Middle and advanced esophageal cancer.
- Normal group: Confirmed as the normal by health checkups.

SUMMARY:
The aim of this study was to detect the whole genome hydroxymethylation of peripheral blood ct DNA in normal population, patients with p0~pI esophageal squamous cell carcinoma and pII~pIV esophageal squamous cell carcinoma by using DNA methylation detection technology. To compare the differences in genomic methylation levels between different groups, to find out the methylolation site system associated with early esophageal squamous cell carcinoma, and to verify the genes related to esophageal squamous cell carcinoma by ctDNA methylolation. Application of basicization in early screening of esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
The aim of this study was to detect the whole genome hydroxymethylation of peripheral blood ct DNA in normal population, patients with p0~pI esophageal squamous cell carcinoma and pII~pIV esophageal squamous cell carcinoma by using DNA methylation detection technology. The differences in genomic methylation levels between different groups were compared to identify the methylolation site system associated with early esophageal squamous cell carcinoma. Then, using the genomic methylolation technique, 5hmC-DNA enrichment was performed on the peripheral venous blood samples of the experimental group before surgery and the peripheral venous blood samples of the control group, respectively, and then the high abundance and high significance were selected. The 5hmC-DNA fragment was verified by PCR amplification. The genes related to esophageal squamous cell carcinoma were verified by ctDNA methylolation. Finally, the methylolation genes related to esophageal squamous cell carcinoma were identified, and the application of DNA methylation in early screening of esophageal squamous cell carcinoma was explored.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of esophageal squamous cell carcinoma by pathological cytology and histology.
2. Clinically judged patients with p0~pIV initial treatment.（1 Variable risk factors are overeating food (habits) and family history. 2 Among all the patients, the ratio of male to female is 3:1, and the age is between 50 and 70 years old. In addition to eating too hot food, other eating habits (such as eating fresh fruits and vegetables, eating preserved food, etc.) are consistent, other factors (such as BMI, smoking, drinking, etc.) as much as possible. 3 In order to rule out the interference of other diseases, each sample needs to be determined to have no history of other diseases (such as neurodegenerative diseases, leukemia).）
3. The normal population comes from the healthy population of Nanfang Hospital Health Center of Southern Medical University.

Exclusion Criteria:

1. Preoperative patients have received relevant treatment, such as radiotherapy and chemotherapy;
2. The subject has other diseases, such as tumors in other parts;
3. Patients do not meet the age;
4. There is no guarantee that other eating habits (such as eating fresh fruits and vegetables, not eating preserved foods) and other factors (such as BMI, smoking, drinking, etc.) are basically the same.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population comes from the Nanfang Hospital of Southern Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Hydroxymethylation level | up to 2 years
  To compare the differences in hydroxymethylation levels among patients in different groups, to identify the hydroxymethylation genes associated with esophageal squamous cell carcinoma, and to verify the genes related to esophageal squamous cell carcinoma by ctDNA hydroxymethylation.

CONTACTS AND LOCATIONS:
Overall Officials: kaican cai, Study Director — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided